CLINICAL TRIAL: NCT05300451
Title: A Phase II Prospective Study Evaluating the Role of Daratumumab in HLA Desensitization Prior to Transplantation
Brief Title: Daratumumab in HLA Desensitization Prior to Transplantation
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Barry A. Boilson (Other)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Barry A. Boilson, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-012885
Record Dates: First submitted 2022-02-08; First posted 2022-03-29 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Transplant
Keywords: Sensitisation; HLA
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLA Desensitization Group (Experimental): Subjects awaiting cardiac transplantation with high levels of circulating Human Leukocyte Antigen (HLA) antibodies will receive daratumumab/hyaluronidase-fihj.
  Interventions: Biological: Daratumumab and hyaluronidase-fihj

INTERVENTIONS:
Biological: Daratumumab and hyaluronidase-fihj — Daratumumab and hyaluronidase-fihj for subcutaneous (under the skin) injection has different dosing and administration instructions compared to daratumumab for intravenous (in the vein) infusion. Daratumumab and hyaluronidase-fihj contains recombinant hyaluronidase, which mimics hyaluronidase, a naturally occurring substance that increases permeability of subcutaneous tissue. This makes it possible for 15 mL containing 1,800 mg of daratumumab to be administered in approximately 3 to 5 minutes. Subjects will receive a 1800mg/30000u injection subcutaneously weekly for a total of 8 doses
  Other Names: DARZALEX FASPRO®

SUMMARY:
The purpose of this study is to learn about how well the drug daratumumab/hyaluronidase-fihj (DARZALEX Faspro™) helps to lower high levels of HLA (Human Leukocyte Antigen) antibodies in a person waiting for a heart transplant.

DETAILED DESCRIPTION:
Daratumumab is an IgG1k, CD38-targeting monoclonal antibody, and the IV formulation was United States Food and Drug Administration (FDA) approved in 2015 for the treatment of multiple myeloma. Daratumumab has not been approved for the indication being studied in this current trial and has been granted investigational new drug (IND) approval by the FDA (IND 157466) for use in this research.

Subjects treated for HLA desensitization will be in the study for 16 weeks. Each subject will receive daratumumab/hyaluronidase-fihj 1800mg/30000u subcutaneously once a week for 8 weeks.

Subjects will have close follow-up for several weeks afterwards with usual testing to monitor for rejection after transplantation. This includes echocardiograms, heart biopsy or MRI and blood tests.

Janssen Biotech, Inc. is providing the daratumumab/hyaluronidase-fihj (DARZALEX Faspro™) for the study.

ELIGIBILITY:
General Inclusion Criteria:

* Absolute neutrophil count > 1,500
* Total bilirubin < 1.5x institutional upper limit normal (ULN)
* AST/ALT < 2. 5 - 3x ULN (Options for patients with liver dysfunction may be available)
* Creatinine clearance > 20 ml/min

Specific Inclusion Criteria [HLA Desensitization Group]

* Calculated PRA (cPRA) greater than 50%.
* Currently actively listed for heart or combined heart and kidney transplantation.
* Negative pregnancy test (if woman of childbearing potential) If able to become pregnant or father a child, agreement to use one of the birth control methods described in this protocol
* Able to provide informed consent

General Exclusion Criteria:

* Prior or current exposure to any of the following: daratumumab or other anti-CD-38 therapies, exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
* Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.
* Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
* Woman who is pregnant or breastfeeding. Participant is: known history of human immunodeficiency virus (HIV); Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative with antibodies to total hepatitis B core antigen [anti-HBc] with or without the presence of hepatitis B surface antibody [anti-HBs]) must be screed using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of HBV vaccination, do not need to be testing for HBV DNA by PCR; Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

Clinically significant cardiac disease, including: myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV); Uncontrolled cardiac arrhythmia

Specific Exclusion Criteria [HLA Desensitization Group]

* Patients listed for combined heart and liver transplantation will be excluded, as our unique experience with combined heart liver transplant (liver placed first), has demonstrated that in those cases high levels of circulating HLA antibodies may not increase the risk of hyperacute rejection.
* Seropositivity for human immunodeficiency virus (HIV)
* Seropositivity for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Seropositivity for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Patients unable to give informed consent will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Effect of daratumumab therapy on human leukocyte antibody (HLA) titers in resistant antibody mediated rejection (AMR) | Sixteen weeks
  Levels of HLA titers by measure of fluorescence intensity levels (MFI) of donor specific antibodies (DSA).
Effect of daratumumab therapy on HLA antibody titers in sensitization (pre-transplant) | Sixteen weeks
  Assessed as calculated panel of reactive antibodies (cPRA) and absolute HLA antibody levels (MFI)

SECONDARY OUTCOMES:
Effect of daratumumab on cardiac contractility in HLA sensitized patients | One month post completion
  As measured by a change in left ventricle (LV) ejection fraction percentage.
Effect of daratumumab on Cardiac Systolic Strain in HLA sensitized patients | One month post completion
  Assessed by echocardiogram and measured by a change in Global LV Longitudinal Peak Systolic Strain percentage, which is the measure of the degree of change in cardiac shape that occurs during systole and diastole.
Effect of daratumumab on Left Ventricular Filling Pressure Ratio in HLA sensitized patients | One month post completion
  Assessed by echocardiogram and measured as a change in the ratio (E/e') between early mitral inflow velocity and mitral annual diastolic velocity.
Effect of daratumumab on Right Ventricular Systolic Pressure (RVSP) in HLA sensitized patients | One month post completion
  Assessed by echocardiogram as a change in approximate pulmonary arterial systolic pressure. Units are mmHg (millimeters of mercury).
Effect of daratumumab on incidence of acute CMR post-transplant in sensitized patients | Time Frame: Weeks 2, 3 and 4 post-transplant
  Evidence of CMR (cellular mediated rejection) based on post-transplant biopsy findings. CMR is scored as follows:
  * Grade 0R: no rejection.
  * Grade 1R, mild: interstitial or perivascular infiltrate (or both) with £1 focus of myocyte damage.
  * Grade 2R, moderate: ³2 foci of infiltrate with associated myocyte damage.
  * Grade 3R, severe: diffuse infiltrate with multifocal myocyte damage, with or without edema, hemorrhage, or vasculitis.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Boilson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials